CLINICAL TRIAL: NCT01906099
Title: Effects of Legume Intake on Cardiovascular Risk Factors Among Adults at Risk for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: legume intake and CVD risks
Record Dates: First submitted 2013-07-09; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- legume enriched diet (Experimental): legume consumption, 4 servings per week, for 6 weeks
  Interventions: Other: nutritional intervention
- healthy dietary recommendations (Active Comparator): no nutritional intervention
  Interventions: Other: life style modification

INTERVENTIONS:
Other: nutritional intervention
  Arms: legume enriched diet
Other: life style modification
  Arms: healthy dietary recommendations

SUMMARY:
This randomized cross-over study was designed to investigate the effects of legume enriched diet consumption on cardiovascular risk factors among first degree relatives of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged more than 30 years
* no history of chronic diseases
* no use of blood glucose lowering drugs be wiling to participate to study

Exclusion Criteria:

* do not follow study protocol
* incidence of chronic diseases during the study
* to start use of blood glucose lowering drugs or to change dose and type of current medications

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose (mg/dl) | 14 weeks
  amounts of FBG

SECONDARY OUTCOMES:
Hemoglobin A1C (%) | 14 weeks
  amounts of HbA1C
Total cholesterol (mg/dl) | 14 weeks
  amounts of TC
Low Density Lipoprotein (mg/dl) | 14 weeks
  amounts of LDL
High Density Lipoprotein (mg/dl) | 14 weeks
  amounts of HDL
Triglyceride (mg/dl) | 14 weeks
  amounts of TG

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran